CLINICAL TRIAL: NCT03777943
Title: Role of the Peritoneal Microenvironment in the Pathogenesis and Spread of Colorectal Carcinomatosis
Acronym: MMT
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Belgian Federation Against Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2017/0784
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cytoreductive surgery (CRS): In patients presenting with colorectal peritoneal carcinomatosis, peritoneal tissue will be sampled during surgery at 4 different locations.
  Interventions: Procedure: Sampling peritoneal tissue

INTERVENTIONS:
Procedure: Sampling peritoneal tissue — Resection specimen will be obtained during CRS from normal peritoneum at a distance, normal peritoneum close to a peritoneal metastasis, miliary peritoneal carcinomatosis, and established peritoneal carcinomatosis.

SUMMARY:
The goal of this project is to investigate the extent and role of mesothelial - mesenchymal transition (MMT) and cancer associated fibroblasts (CAFs) in the pathogenesis of colorectal peritoneal carcinomatosis (PC).

ELIGIBILITY:
Inclusion Criteria:

• Patients presenting with colorectal peritoneal carcinomatosis

Exclusion Criteria:

* Pregnancy or breast feeding
* Psychiatric pathology capable of affecting comprehension and judgment faculty
* HIPEC (hyperthermic intraperitoneal chemotherapy) or PIPAC (pressurized intraperitoneal aerosol chemotherapy) in the past
* Abdominal radiation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with colorectal peritoneal carcinomatosis
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Immunohistochemistry (IHC) analysis | Within 6 months after collection of the samples
  Extensive IHC analysis will be performed including CD44, integrins, ICAM-1, hyaluronate, and VCAM-1 (adhesion molecules); calretinin, mesothelin, WT1, cytokeratins and E-cadherin (mesothelial markers); α-SMA, FAP and podoplanin (CAF specific markers); PDGF, VEGF and EDGF (angiogenesis related markers)

SECONDARY OUTCOMES:
Intra-tumoral versus peritoneal vascularity | Within 6 months after collection of the samples
  Vacularity will be assed using chalkley counts
Laser capture microdisssection (LCM) followed by gene expression analysis | Within 12 months after collection of the samples
  Different cell types (mesothelial cells, submesothelial resident fibroblasts, CAFs) will be isolated using LCM, followed by gene expression analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No